CLINICAL TRIAL: NCT06030518
Title: Feasibility and Acceptability of Robot-controlled Magnet-Assisted Capsule Endoscopy Compared to Conventional Endoscopy of the Upper Gastrointestinal Tract in Children
Brief Title: Robot-controlled Magnet-Assisted Capsule Endoscopy
Acronym: MACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH-2497
Record Dates: First submitted 2022-09-21; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-06

CONDITIONS: Abdominal Pain; Upper Gastrointestinal Symptoms
Keywords: Upper GI endoscopy
MeSH Terms: conditions — Abdominal Pain | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient undergoing upper Gi endoscopy (Experimental): Children attending Sheffield Childrens' Hospital Gastroenterology out-patients departments between the ages of 11-16 years of age who require OGD to investigate abdominal pain or discomfort will be invited to take part in the study.
  Interventions
  The study will begin when capsule endoscopy is performed by a Clinical Research Fellow at the Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS Trust.
  Interventions: Diagnostic Test: Magnet Assisted Capsule Endoscopy

INTERVENTIONS:
Diagnostic Test: Magnet Assisted Capsule Endoscopy — Procedures will be performed in the morning after an overnight fast. Patients wear a belt containing sensors and a data recorder. The patient will be asked to drink 500-1000ml (containing 80mg simethicone; volume depending on tolerance) immediately before swallowing the capsule. Gastric examination will proceed as previously described for a robot-controlled magnetic assisted capsule endoscopy. The whole procedure is anticipated to take 30-60 minutes. The patient will be discharged from hospital on completion of gastric examination but if clinically indicated will wear the belt for small bowel capsule study for eight hours to allow small bowel examination before detaching the equipment and returning it the following day. On completion of examination, the patient will be asked to complete a questionnaire about their capsule endoscopy experience. The full study (upper GI tract and small bowel) will then be downloaded onto the computer for formal reading and reporting.

SUMMARY:
Examination of the upper gastrointestinal tract (oesophagus, stomach and duodenum) involves passing a flexible tubular endoscope through the mouth into the stomach. It is commonly performed to identify the cause of abdominal pain, indigestion, diarrhoea and anaemia. As it is an invasive and uncomfortable test, it is usually performed under general anaesthetic in children. However, children and their parents worry about the nature of the procedure which does incur a small risk of both the anaesthetic and the endoscopy.

A capsule endoscope is a large pill-sized device containing a battery powered camera which can be swallowed. It was first devised to examine the small bowel (which begins with the duodenum and ends in the colon or large bowel) which is difficult to reach with conventional endoscopes and has been used in children aged over eight years since at least 2005. It is extremely well tolerated. However, it does not provide a comprehensive view of the whole surface area of the stomach which has a convoluted shape, large volume and is collapsed in the fasted state.

Recent research in adults shows that a capsule can be steered around a water-filled stomach using two joysticks to control the polarity and distance of an external robot magnet from the patient. This is much better tolerated and appears to be almost as good a diagnostic tool as conventional endoscopy. It has yet to be studied in children. We intend to compare patient acceptability of capsule endoscopy and gastroscopy and see if it is cost effective.

DETAILED DESCRIPTION:
A capsule endoscope is a swallowable pill camera (26x11mm) which images the GI tract as it passes through under the action of peristalsis. It is a non-invasive test which does not require sedation or general anaesthesia. It was originally designed to image the small bowel, which is inaccessible to conventional endoscopy, and was subsequently adapted for use in the colon by the addition of a second camera (one at each end of the device) and a higher frame acquisition rate. The unusual configuration of the oesophagus, stomach and duodenum, the capacious and non-uniform shape of the stomach and the fact that it is collapsed in the fasted state presented barriers to extending examination to the upper gastrointestinal tract. However, recent studies in adult patients with anaemia, suspected upper gastrointestinal bleeding and dyspepsia suggest that capsules which are steered around the stomach in swallowed water using external magnets achieve comparable diagnostic yields to OGD. Control is achieved using a magnet suspended above the patient who is recumbent on an examination couch. The examiner manipulates two joysticks to alter the polarity of the magnet and its distance from the patient to steer the capsule around whilst conducting a live inspection of the stomach on a computer monitor. An additional benefit is that the small bowel can be examined following passage of the capsule through the stomach, which further improves the diagnostic yield.

Studies in the adult population suggest that capsule endoscopy of small bowel, colon and upper gastrointestinal tract is much better tolerated than conventional (invasive) endoscopy. Capsule endoscopy is a recommended investigation for suspected small bowel disease in children over the age of two years. Young children may need a small bowel capsule to be delivered endoscopically, but 85- 90% of children of over eight years of age are able to swallow it with water and 82% of 28 children expressed a preference for capsule endoscopy over conventional endoscopy (done under deep sedation or general anaesthesia) in one study. Magnetically controlled upper GI capsule endoscopy may offer a better tolerated, more acceptable alternative to OGD in children. Secondly, the ability to provide upper GI imaging without general anaesthetic may be a more cost-effective approach. Finally, such a non-invasive diagnostic tool could be used as a near-patient test, performed in the patients' community rather than an acute hospital setting.

This study proposes comparing patient acceptability and cost-effectiveness of capsule endoscopy compared to OGD in children.

The joystick-controlled robot magnet used for upper GI capsule endoscopy is on the Clinical Investigation Unit at the Royal Hallamshire Hospital, Sheffield, where it is being used in clinical trials and routine clinical practice in adults. It was the first of four systems (two in France and one in Hungary) to be installed outside of China.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal pain requiring investigation by OGD
* Participant must be willing to undergo both procedures (i.e. ingestion of the capsule and standard of care Oesophago-gastro duodenoscopy (OGD)
* Age 11-16 years inclusive

Exclusion Criteria:

* Dysphagia
* Inability to swallow capsule
* Small bowel stricture
* Disease associated with small bowel stricturing (Crohn's disease, previous small bowel surgery, previous abdominal or pelvic radiation therapy, long term daily (>6 months) non-steroidal anti-inflammatory drug consumption)
* Pacemaker or other implantable electrical cardiac or neurological device
* Unable to speak English
* Participants who are pregnant or who have implantable electronic devices cannot take part in the study. Depending on their age and pubertal status the female patients will be offered a pregnancy test prior to any examinations. Capsule endoscopy is not advised during pregnancy.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of upper GI capsule endoscopy | One year
  Compare acceptability of upper GI capsule endoscopy and OGD in children using UPC questionnaire.

SECONDARY OUTCOMES:
Diagnostic Yield | One year
  Compare diagnostic yield of upper GI capsule endoscopy and OGD in children
Prevalence of small bowel pathology | One year
  Determine the prevalence of small bowel pathology as a cause for abdominal pain in children.

CONTACTS AND LOCATIONS:
Overall Officials: Shishu Sharma, Study Chair — Sheffield Childrens NHS FT
Locations (1):
- Sheffield Childrens NHS FT, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No